CLINICAL TRIAL: NCT05443555
Title: Gabapentin to Reduce Alcohol and Improve Viral Load Suppression - Promoting "Treatment as Prevention"
Brief Title: Gabapentin to Reduce Alcohol and Improve Viral Load Suppression
Acronym: GRAIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-42904; R01AA030460 (NIH)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: HIV; Heavy Drinking
Keywords: Uganda; Alcohol Use; ART; HIV; Gabapentin
MeSH Terms: conditions — Alcohol Drinking | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention: Gabapentin (Active Comparator): Participants randomized to the intervention group will receive active gabapentin for 3 months and brief (5-minute) evidence-based counseling for alcohol use.
  Interventions: Drug: Gabapentin
- Control: Placebo (Placebo Comparator): Participants randomized to the control group will receive placebo capsules, identical in appearance to gabapentin, and the same brief (5-minute) one-time evidence-based counseling for alcohol use as the intervention group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Dosing will be titrated up over 3 weeks, starting with a daily dose of 300mg (1 capsule/day) in week 1, followed by a daily dose of 900mg (3 capsules/day) in week 2, up to a target daily dose of 1800mg (6 capsules/day) in week 3. The target dose of 1800mg per day will be sustained from weeks 3 through day 4 of week 12. Then, dose will be tapered down to 900mg in days 5-7 of week 12, and medication will be discontinued at the end of week 12.
  Arms: Intervention: Gabapentin
Drug: Placebo — Participants randomized to this group will receive a placebo medication for 3 months and will be instructed to follow the same pill regimen as the intervention arm.
  Arms: Control: Placebo

SUMMARY:
GRAIL is a Randomized Controlled Trial (RCT) among 300 HIV-positive persons with heavy alcohol consumption (by NIAAA definition) who have had detectable HIV viral load (HVL) at least 6 months after their HIV diagnosis. This trial aims to test the efficacy of gabapentin versus placebo to achieve undetectable HVL and assess the impact of gabapentin compared to placebo on alcohol consumption, pain severity, ART adherence, and engagement in HIV care. HIV viral load will be assessed at 3 (primary), 6 and 12 months via laboratory test. Eligible participants will be randomly assigned into one of two study arms: 1) gabapentin (1800mg/day target dose) for 3 months vs. 2) placebo for 3 months. All participants will receive evidence-based counseling for alcohol and either an active medication or placebo.

DETAILED DESCRIPTION:
Ending the HIV epidemic requires achieving HIV viral load (HVL) suppression (i.e., undetectable viral load) for key populations. Unhealthy alcohol use by people with HIV (PWH) is a barrier to reaching HVL suppression at multiple stages of the HIV care cascade. Alcohol use is common among PWH and results in lower antiretroviral therapy (ART) adherence and HVL suppression, mitigating the effectiveness of Treatment as Prevention (TasP), a key strategy for preventing HIV transmission. Treating alcohol use is therefore a mechanism to support PWH with unhealthy alcohol use along the HIV care cascade (e.g., ART initiation, retention in care, medication adherence, and HVL suppression).

The investigators propose the Gabapentin to Reduce Alcohol and Improve Viral Load Suppression (GRAIL) trial to test the efficacy of gabapentin vs. placebo on achieving viral load suppression among PWH. The study population will be heavy drinkers with a detectable viral load at least 6 months after their HIV diagnosis. The rationale for this trial is that effective pharmacological alcohol treatment will help PWH with heavy alcohol use who have a known HIV diagnosis for at least 6 months to successfully engage in HIV care. The overarching strategy to achieve TasP is that gabapentin will reduce heavy alcohol use, thereby increasing HIV care engagement, ART use and adherence while decreasing pain, all of which ultimately promote viral load suppression.

GRAIL is a randomized, double-blinded, placebo-controlled clinical trial that will evaluate the efficacy of gabapentin in promoting HVL suppression via reducing alcohol use among PWH but not virally suppressed (i.e., The study population will be heavy drinkers with a detectable viral load for 6 months or more after their HIV diagnosis). Participants will be randomized 1:1 to receive either gabapentin (1800mg/day target dose) or placebo for 3 months; both arms will employ a brief intervention to reduce alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Having an HIV diagnosis for at least 6 months
* Current (within 2 months) detectable HIV viral load at least 6 months after HIV diagnosis
* Positive EtG urine test
* Able and willing to comply with all study protocols and procedures
* Living within 2 hours travel time of the study site

Exclusion Criteria:

* Not fluent in English or Runyankole
* Cognitive impairment resulting in inability to provide informed consent based on research assessor (RA) assessment
* Pregnancy, planning to become pregnant in next 3 months, or breast feeding
* Taking gabapentin/pregabalin in past 30 days
* Taking any medication for alcohol use disorder
* Enrolled in another HIV research study seeking viral load suppression
* Known hypersensitivity to gabapentin
* Unstable psychiatric illness (i.e., answered yes to any of the following: past three month active hallucinations; mental health symptoms prompting a visit to the emergency department (ED) or hospital; mental health medication changes due to worsening symptoms; presence of suicidal ideations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with undetectable HIV viral load | 3 months post randomization
  Assessed by study test

SECONDARY OUTCOMES:
Number of participants with undetectable HIV viral load | 6 months post randomization
  Assessed by study test
Number of participants with undetectable HIV viral load | 12 months post randomization
  Assessed by study test

OTHER OUTCOMES:
Number of heavy drinking days in the past month | 3, 6, and 12 months post randomization
  Assessed by self-report using the Timeline Followback method
Number of participants with heavy alcohol consumption defined as Phosphatidylethanol (PEth) ≥50 ng/mL | 3, 6, and 12 months post randomization
  Assessed by study test
Adherence to ART | 3, 6, and 12 months post randomization
  Measured by participants' drawing a line on a Visual Analog Scale, which ranges from 0 to 100. ≥80% indicates adherence to ART.
Percentage of ART pills taken | 3, 6, and 12 months post randomization
  Assessed by self-report
Change in pain severity from baseline to follow-up | 3, 6, and 12 months post randomization
  Assessed by Brief Pain Inventory with a range of scores from 0 (none) to 10 (high) where lower scores are favorable.
Engagement in HIV care | 3, 6, and 12 months post randomization
  Defined as ≥ 1 HIV visit in the past 3 months assessed by medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD MA MPH, Principal Investigator — Boston University; Karsten Lunze, MD MPH DrPH, Principal Investigator — Boston University
Locations (1):
- Mbarara Regional Referral Hospital (MRRH): Immune Suppression Syndrome HIV, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Truong V, Kekibiina A, Muyindike W, Gnatienko N, Tsui JI, Emenyonu NI, Cheng DM, Hahn J, Allison O, Bullard MJ, Lunze K, Samet JH. Gabapentin to achieve HIV viral load suppression in people with risky drinking in Mbarara, Uganda: study protocol for a randomized, double-blinded, placebo-controlled trial (GRAIL). Res Sq [Preprint]. 2025 Oct 15:rs.3.rs-6856284. doi: 10.21203/rs.3.rs-6856284/v1. PMID 41282191